CLINICAL TRIAL: NCT06292611
Title: Clinical Evaluation of a Powered Toothbrush in Tooth Whitening Via Extrinsic Stain Removal
Brief Title: Two Week Cumulative Extrinsic Stain Removal of a Battery-powered Toothbrush and a Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST-23-U35
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Battery operated toothbrush (Active Comparator): Battery operated toothbrush
  Interventions: Device: Battery operated toothbrush
- Manual toothbrush (Active Comparator): Manual toothbrush
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Battery operated toothbrush — Device on extrinsic stain removal efficacy
  Arms: Battery operated toothbrush
Device: Manual toothbrush — Device on extrinsic stain removal efficacy
  Arms: Manual toothbrush

SUMMARY:
To evaluate and compare the extrinsic stain removal efficacy of a battery-powered toothbrush and a manual toothbrush following two weeks of brushing.

DETAILED DESCRIPTION:
This is a two week, examiner blinded, randomized, parallel group, IRB-approved research study evaluating the extrinsic stain removal efficacy of a new battery-operated toothbrush and a marketed manual toothbrush. This study will accept up to 110 subjects, 18-65 years of age, in anticipation that 50 subjects per treatment group will complete the study. Qualified subjects with sufficient extrinsic stain, according to Macpherson Modified Lobene Stain Index (MLSI) will be randomly assigned to one of two treatment groups.

Subjects will brush with the assigned toothbrush and toothpaste provided for timed brushing twice a day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 65, ambulatory and in good general health as determined by the Study Examiner, based upon clinical observation and the Medical/Dental History;
2. Be able to understand and sign the Informed Consent, complete a Medical History form, understand and comply with all study directions, and be available for all exam periods;
3. Present with adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of oral neglect) and continue to meet the inclusion criteria and not fall into the categories of exclusion during the period of the study;
4. Have at least 16 natural teeth in a good state of repair and at least 8 of the 12 anterior teeth free from full crowns or extensive restorations;
5. Have a mean Macpherson Modified Lobene Stain Index (MLSI) score of ≥ 1.5 on the labial surfaces of at least 8 of 12 anterior teeth;
6. Have had a dental prophylaxis within the past 18 months, but not within the past 3 months;
7. Agree to refrain from using all oral care products (other dentifrices and toothbrushes, dental floss, and mouth rinses) other than their assigned products for the duration of the study.
8. Agree to comply with the conditions and schedule of the study; and
9. Approximately 50% of study participants will be regular power brush users, with the remaining 50% of study participants regular manual brush users.

Exclusion Criteria:

1. Have a history of serious medical conditions or transmittable diseases including but not limited to COVID-19, active hepatitis, heart irregularities, conditions requiring pre-medication for dental procedures, rheumatic heart disease, untreated diabetes mellitus, cirrhosis, leukemia, phenylketonuria, renal disease, sarcoidosis, tuberculosis, bleeding disorder, vascular disease, AIDS, history of drug allergies or idiosyncrasies, or any other medical condition that may preclude successful participation in the trial, at the discretion of the Study Examiner;
2. Have had prior significant adverse effects following use of oral hygiene products;
3. Have the presence of orthodontic bands, retainers, fixed appliances, large restorations, or removable partial dentures, which may interfere with clinical assessments of the evaluable teeth;
4. Show evidence of neglected dental health in need of prompt professional attention (i.e. gross calculus deposits or rampant caries), significant oral soft tissue pathology, systemically-related gingival enlargement, generalized recession, tissue damage due to ill-fitting appliances or restorations or extreme crowding or overlapping of teeth;
5. Have moderate/advanced periodontitis (ADA Class III or IV), e.g. more than two teeth with periodontal pockets >4 mm as evidenced by purulent exudate, tooth mobility, and other signs indicating that the integrity of the data collected might be compromised;
6. Have medication therapy that is current and ongoing or within the past 4 weeks, which might interfere with the outcome of the study by affecting oral tissue condition, salivation, or stain formation (particularly chronic long-term medication therapy);
7. Are nursing (breast-feeding) or pregnant;
8. Present at baseline with any reported sensory reactions, observed gum irritation or any condition that would interfere with subsequent clinical assessments, or subjects with a history of allergy to oral care products, severe oral cavity sensitivity, or excessive oral irritation;
9. Have participated in tooth bleaching or whitening dentifrice trials within the last three months; and
10. Have had professional or at-home bleaching during the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Extrinsic Stain | 2 weeks
  Macpherson Modification of the Lobene Stain Index (MLSI)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Study Director — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No